CLINICAL TRIAL: NCT06109389
Title: The Efficacy of Intravenous Lidocaine Infusion in Chronic Unilateral Migraine Headache Clinical and Laboratory Assessment .Aprospective Randomized Double Blind Controlled Study
Brief Title: The Efficacy Of Lidocaine Infusion IN Chronic Unilateral Migraine Headache
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E/C.S/N.T71/2023
Record Dates: First submitted 2023-10-11; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Chronic Migraine, Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- infusion of saline (Experimental): infusion saline for 4 successive weeks once weekly over 45 min
  Interventions: Drug: Lidocaine IV
- lidocaine infusion (Active Comparator): infusion of lidocaine 3 mg per kg for 2 successive weeks then 4 mg per kg for 2 successive weeks
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: Lidocaine IV — LIDOCAINE INFUSION STARTED 3 MG PER KG FOR 2 SUCCESSIVE WEEKS ,THEN 4 MG PER KG FOR ANOTHER 2 WEEKS .ONCE WEEKLY,other group saline infusion once weekly for 4 successive weeks
  Other Names: Saline infusion once weekly for 4 successive weeks

SUMMARY:
STUDY THE EFFICACY OF INTRAVENOUS LIDOCAINE INFUSION ON PATIENTS WITH CHRONICUNILATERAL MIGRAINE HEADACHE ..NO OF PATIENTS 80..WILLBE DIVIDED INTO 2 GROUPS..FIRST WILL RECEIVE MEDICAL TREATMENT PLUS LIDOCAINE INFUSION ONCE WEEKLY FOR 4 SUCCESIVE WEEKS ,OTHER WILL RECEIVE MEDICAL TREATMENT PLUS SALINE INFUSION SAME REGIMNE,FOLLOW UP USING MONTHLY MIGRAINE DAYS,VAS SCORE,MIDAS SCORE,QUALITY OF LIFE QUESTIONAIRE,PRE AND POST MEASUREMENT OF CALCITONIN GENE RELATED PEPTIDE

DETAILED DESCRIPTION:
Group A will receive medical treatment for migraine plus normal saline infusion,Group B will receive medical treatment plus lidocaine infusion at dose from 3 to 4 mg per kg,computer generated random number will be used to identify the selected blocks and give the sequence of patients allocation,guarantee equal random in each group a set of permuted blocks will be generated. Each block has 4 differently ordered treatment assignments.Block 1 (AABB),Block2(ABAB),Block3(BABA),Block 4(ABBA),Block5(BAAB),Block 6(BBAA).

ELIGIBILITY:
Inclusion Criteria:

* Age (18-55) years for both genders.
* Patients with chronic unilateral migraine headache for at least (3) month with VASscore more than (4).
* Patient who failed to respond to conservative treatment as medical treatment algorithm including at least tow preventive trials.

Excusion criteria:

* patient with disabling chronic disease or psychiatric illness
* unstable cardiac arrhythmia
* patient refusal red flags

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Monthly Migraine Days | 3 Month
  Number of Migraine Attacks Per Month More or less than (15) for chronicity
Verbal analogue scale for pain | 3 month
  verbal analogue scale for pain from( 0) to( 10) as( 0) no pain( 10) severe pain untolerable

SECONDARY OUTCOMES:
Migraine attack duration | 3 Month
  Duration of each attack from (4) hours to (72) hours
Calcitonin Gene Related Peptide Biomarker. | 3 Month
  Measurement of CGRP before and after( 1) month from first infusion treatment
Migraine Specific Quality Of Life Questionaire | 3 Month
  14 questions ,each one measured from ( 1) never affect to(6) always affect ,answers summed for all questions value is obtained
Migraine Disability Assessment Questionaire | 3 Month
  (0) Absent of disability,(270) Extremely severe disability,more than (21) severe disability

CONTACTS AND LOCATIONS:
Overall Officials: Sahar ah El karadawy, phd, Study Director — Medical Research I nstitute
Locations (1):
- Alexandria University,Medical Research Institute, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data and results will be available to share of other researches after completion
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 to 9 month

REFERENCES:
- [Result] Aggarwal M, Puri V, Puri S. Serotonin and CGRP in migraine. Ann Neurosci. 2012 Apr;19(2):88-94. doi: 10.5214/ans.0972.7531.12190210. PMID 25205974
- [Result] Al Ghadeer HA, AlSalman SA, Albaqshi FM, Alsuliman SR, Alsowailem FA, Albusror HA, AlAbdi ZI, Alwabari EM, Alturaifi ZA, AlHajji AM. Quality of Life and Disability Among Migraine Patients: A Single-Center Study in AlAhsa, Saudi Arabia. Cureus. 2021 Nov 2;13(11):e19210. doi: 10.7759/cureus.19210. eCollection 2021 Nov. PMID 34873540
- [Result] Andreou AP, Edvinsson L. Mechanisms of migraine as a chronic evolutive condition. J Headache Pain. 2019 Dec 23;20(1):117. doi: 10.1186/s10194-019-1066-0. PMID 31870279
- [Result] Eigenbrodt AK, Ashina H, Khan S, Diener HC, Mitsikostas DD, Sinclair AJ, Pozo-Rosich P, Martelletti P, Ducros A, Lanteri-Minet M, Braschinsky M, Del Rio MS, Daniel O, Ozge A, Mammadbayli A, Arons M, Skorobogatykh K, Romanenko V, Terwindt GM, Paemeleire K, Sacco S, Reuter U, Lampl C, Schytz HW, Katsarava Z, Steiner TJ, Ashina M. Diagnosis and management of migraine in ten steps. Nat Rev Neurol. 2021 Aug;17(8):501-514. doi: 10.1038/s41582-021-00509-5. Epub 2021 Jun 18. PMID 34145431
- [Result] Di Tanna GL, Porter JK, Lipton RB, Brennan A, Palmer S, Hatswell AJ, Sapra S, Villa G. Migraine day frequency in migraine prevention: longitudinal modelling approaches. BMC Med Res Methodol. 2019 Jan 23;19(1):20. doi: 10.1186/s12874-019-0664-5. PMID 30674285
- [Result] Hand PJ, Stark RJ. Intravenous lignocaine infusions for severe chronic daily headache. Med J Aust. 2000 Feb 21;172(4):157-9. doi: 10.5694/j.1326-5377.2000.tb125538.x. PMID 10772585
- [Result] Katsarava Z, Buse DC, Manack AN, Lipton RB. Defining the differences between episodic migraine and chronic migraine. Curr Pain Headache Rep. 2012 Feb;16(1):86-92. doi: 10.1007/s11916-011-0233-z. PMID 22083262
- [Result] Lipton RB, Diamond S, Reed M, Diamond ML, Stewart WF. Migraine diagnosis and treatment: results from the American Migraine Study II. Headache. 2001 Jul-Aug;41(7):638-45. doi: 10.1046/j.1526-4610.2001.041007638.x. PMID 11554951
- [Result] Mungoven TJ, Henderson LA, Meylakh N. Chronic Migraine Pathophysiology and Treatment: A Review of Current Perspectives. Front Pain Res (Lausanne). 2021 Aug 25;2:705276. doi: 10.3389/fpain.2021.705276. eCollection 2021. PMID 35295486
- [Result] Schoenen J, Timmermans G, Nonis R, Manise M, Fumal A, Gerard P. Erenumab for Migraine Prevention in a 1-Year Compassionate Use Program: Efficacy, Tolerability, and Differences Between Clinical Phenotypes. Front Neurol. 2021 Dec 10;12:805334. doi: 10.3389/fneur.2021.805334. eCollection 2021. PMID 34956071
- [Result] Myles PS, Urquhart N. The linearity of the visual analogue scale in patients with severe acute pain. Anaesth Intensive Care. 2005 Feb;33(1):54-8. doi: 10.1177/0310057X0503300108. PMID 15957691
- [Result] Schwenk ES, Walter A, Torjman MC, Mukhtar S, Patel HT, Nardone B, Sun G, Thota B, Lauritsen CG, Silberstein SD. Lidocaine infusions for refractory chronic migraine: a retrospective analysis. Reg Anesth Pain Med. 2022 Jul;47(7):408-413. doi: 10.1136/rapm-2021-103180. PMID 35609890
- [Result] Fink R. Pain assessment: the cornerstone to optimal pain management. Proc (Bayl Univ Med Cent). 2000 Jul;13(3):236-9. doi: 10.1080/08998280.2000.11927681. PMID 16389388